CLINICAL TRIAL: NCT03446144
Title: A Phase 2, Placebo-Controlled, Double-Masked Study to Assess Safety and Efficacy of ISIS 696844, an Antisense Inhibitor of Complement Factor B, in Patients With Geographic Atrophy Secondary (GA) to Age-Related Macular Degeneration (AMD)
Brief Title: Safety and Efficacy of IONIS-FB-Lrx in up to 120 Patients 55 and Older With Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration (AMD)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objective change, no safety or efficacy concerns
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISIS 696844-CS3
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Geographic Atrophy; Age Related Macular Degeneration
Keywords: Geographic Atrophy; Age Related Macular Degeneration; IONIS-FB-Lrx; Complement Factor B
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Masked
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IONIS-FB-Lrx (Experimental)
  Interventions: Drug: IONIS-FB-Lrx
- Placebo (sterile saline 0.9%) (Placebo Comparator)
  Interventions: Drug: Placebo (sterline saline 0.9%)

INTERVENTIONS:
Drug: IONIS-FB-Lrx — Single Dose of IONIS-FB-Lrx administered once weekly for weeks 1-3, and every other week or less frequently until week 70
  Arms: IONIS-FB-Lrx
Drug: Placebo (sterline saline 0.9%) — Calculated volume to match active comparator. Administered subcutaneously weekly for weeks 1-3, and every other week or less frequently until week 70
  Arms: Placebo (sterile saline 0.9%)

SUMMARY:
The purpose of this study is to assess the Safety and Efficacy of IONIS-FB-Lrx for up to 120 patients with Geographic Atrophy secondary to Age Related Macular Degeneration

DETAILED DESCRIPTION:
This study will assess changes in complement factor B over a 69-week treatment period in a patient population 55 and older with well-demarcated Geographic Atrophy secondary to Age Related Macular Degeneration

ELIGIBILITY:
Key Inclusion Criteria:

1. Must have given written informed consent and be able to comply with study requirements
2. Females must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal. Males must be surgically sterile or, if engaged in sexual relations with a female of child bearing potential, the subject must be using an acceptable contraceptive method from the time of signing the informed consent form until at least a period of 13 weeks after the last dose of Study Drug (ISIS 696844 or placebo)
3. Well-demarcated Geographic Atrophy due to Age Related Macular Degeneration

Key Exclusion Criteria:

1. Clinically-significant abnormalities in medical history
2. Diagnosis of primary or secondary immunodeficiencies of B lymphocyte function, splenectomy, glomerulonephritis or history of recurrent meningococcal disease
3. Diabetes mellitus or thyroid disease unless well controlled for a period of at least 3 months
4. Clinically-significant abnormalities in screening laboratory values
5. Unwillingness to be administered, or history of a serious reaction to protocol required vaccines
6. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
7. History or presence of a disease other than AMD in study eye

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of IONIS-FB-Lrx | Up to 74 weeks
  The Efficacy of IONIS-FB-Lrx will be measured by the percent change in plasma complement factor B level

SECONDARY OUTCOMES:
Incidence and severity of adverse events that are related to treatment with IONIS-FB-Lrx | Up to 86 weeks
  The safety and tolerability of IONIS-FB-Lrx will be assessed by determining the incidence and severity of adverse events that are related to treatment with IONIS-FB-Lrx
Proportion of patients in each treatment group achieving a >50% reduction of plasma complement factor B | Up to 74 weeks
  Proportion of patients in each treatment group achieving a >50% reduction of plasma complement factor B from Baseline to Post-Treatment
Effect of IONIS-FB-Lrx on the rate of change of the area of GA secondary to AMD | Up to 74 weeks
  Effect of IONIS-FB-Lrx on the rate of change of the area of GA secondary to AMD as measured by Fundus Autofluorescence from Baseline to Post-Treatment
Effect of factor B reduction on other components of the complement pathways in AMD patients | Up to 74 weeks
  Effect of factor B reduction on other components of the complement pathways such as AH50, CH50 and Bb in AMD patients from Baseline to Post-Treatment

CONTACTS AND LOCATIONS:
Locations (36):
- United States (23):
  - IONIS Investigative Site, Phoenix, Arizona
  - IONIS Investigational Site, Beverly Hills, California
  - IONIS Investigative Site, Encino, California
  - IONIS Investigative Site, Irvine, California
  - IONIS Investigational Site, Mountain View, California
  - IONIS Investigational Site, Santa Barbara, California
  - IONIS Investigative Site, Clearwater, Florida
  - IONIS Investigational Site, Tampa, Florida
  - IONIS Investigational Site, Augusta, Georgia
  - IONIS Investigational Site, Leawood, Kansas
  - IONIS Investigative Site, Chesterfield, Missouri
  - IONIS Investigative Site, New York, New York
  - IONIS Investigative Site, Philadelphia, Pennsylvania
  - IONIS Investigative Site, Pittsburgh, Pennsylvania
  - IONIS Investigational Site, Ladson, South Carolina
  - IONIS Investigative Site, Rapid City, South Dakota
  - IONIS Investigative Site, Arlington, Texas
  - IONIS Investigational Site, Austin, Texas
  - IONIS Investigative Site, Dallas, Texas
  - IONIS Investigative Site, Houston, Texas
  - IONIS Investigative Site, McAllen, Texas
  - IONIS Investigative Site, San Antonio, Texas
  - IONIS Investigative Site, The Woodlands, Texas
- Australia (12):
  - Eye Clinic Albury Wodonga, Albury, New South Wales
  - IONIS Investigational Site, Liverpool, New South Wales
  - Marsden Eye Specialists, Paramatta, New South Wales
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic Day Surgery, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria
  - Retinology Institute, Glen Iris, Victoria
  - Eye Surgery Associates, Malvern, Victoria
  - Eye Surgery Associates, Parkville, Victoria
  - Lions Eye Institute, Nedlands, Western Australia
- Auckland Eye, Auckland, New Zealand